CLINICAL TRIAL: NCT04029155
Title: Conventional vs Ultrathin Bronchoscopy With Transbronchial Needle Aspiration for the Diagnosis of Peripheral Pulmonary Lesions: a Randomized Controlled Trial
Brief Title: Conventional vs Ultrathin Bronchoscopy for Peripheral Pulmonary Lesions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Stefano Gasparini (Other)
Responsible Party: Sponsor-Investigator, Stefano Gasparini, Professor, Università Politecnica delle Marche
Organization: Università Politecnica delle Marche (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: UTB2019
Record Dates: First submitted 2019-07-18; First posted 2019-07-23 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Lung Cancer
Keywords: peripheral pulmonary nodules; ultrathin bronchoscope; transbronchial needle aspiration
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TBNA with Conventional bronchoscope (Active Comparator): patients in this arm will undergo bronchoscopy by a conventional probe
  Interventions: Device: Lung biopsy
- TBNA with a Ultrathin bronchoscope (Experimental): Patients in this arm will undergo bronchoscopy by a ultra thin probe
  Interventions: Device: Lung biopsy

INTERVENTIONS:
Device: Lung biopsy — Transbronchial Needle Aspiration performed via a ultra thin bronchoscope

SUMMARY:
This study's purpose is to evaluate whether the use of an ultra-thin bronchoscope can improve sensitivity and diagnostic yield in peripheral pulmonary nodules. The ultra-thin probe is expected to reach further bronchi and allow to reach peripheral lesions. Moreover, the ability to identify molecular pattern of lung cancer is essential nowadays, and it will be therefore evaluated.

DETAILED DESCRIPTION:
142 patients with at least one peripheral pulmonary nodule will be enrolled. They will underwent randomization in 2 arms: patients in the first arm will undergo transbronchial needle aspiration with a conventional bronchoscope patients in the second arm will undergo transbronchial needle aspiration with a ultra-thin bronchoscope. Every bronchoscopy will be performed by the same operator and will contemplate 3 passes for each nodule, followed by Rapid On-Site Evaluation (ROSE) assessed by a dedicated cytologist. If the cytological on-site evaluation is negative in patients in the first arm, they will be shifted to the second arm. Histological and molecular diagnosis will be assessed by a dedicated pathologist. Data will be collected and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18years;
* presence of at least one peripheral pulmonary lesion ≤ 3 cm on CT scan;
* ability to give an informed consent.

Exclusion Criteria:

* coagulopathy or bleeding diathesis that cannot be corrected;
* severe refractory hypoxemia;
* unstable hemodynamic status;
* inability to give an informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2022-07-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Assess if sensitivity is higher in the "ultrathin" arm than in the "conventional" arm | through study completion, an average of 6 months
  percentage

SECONDARY OUTCOMES:
Assess if diagnostic yield is higher in the "ultrathin" arm than in the "conventional" arm | through study completion, an average of 6 months
  percentage

OTHER OUTCOMES:
Assess if sensitivity is similar in both arms | through study completion, an average of 6 months
  percentage

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Haponik EF, Shure D. Underutilization of transbronchial needle aspiration: experiences of current pulmonary fellows. Chest. 1997 Jul;112(1):251-3. doi: 10.1378/chest.112.1.251. PMID 9228384
- [Background] Harrow EM, Abi-Saleh W, Blum J, Harkin T, Gasparini S, Addrizzo-Harris DJ, Arroliga AC, Wight G, Mehta AC. The utility of transbronchial needle aspiration in the staging of bronchogenic carcinoma. Am J Respir Crit Care Med. 2000 Feb;161(2 Pt 1):601-7. doi: 10.1164/ajrccm.161.2.9902040. PMID 10673206
- [Background] Gasparini S, Silvestri GA. Usefulness of transbronchial needle aspiration in evaluating patients with lung cancer. Thorax. 2005 Nov;60(11):890-1. doi: 10.1136/thx.2005.048728. No abstract available. PMID 16263944
- [Background] Patelli M, Lazzari Agli L, Poletti V, Trisolini R, Cancellieri A, Lacava N, Falcone F, Boaron M. Role of fiberscopic transbronchial needle aspiration in the staging of N2 disease due to non-small cell lung cancer. Ann Thorac Surg. 2002 Feb;73(2):407-11. doi: 10.1016/s0003-4975(01)03447-6. PMID 11845850
- [Background] Trisolini R, Tinelli C, Cancellieri A, Paioli D, Alifano M, Boaron M, Patelli M. Transbronchial needle aspiration in sarcoidosis: yield and predictors of a positive aspirate. J Thorac Cardiovasc Surg. 2008 Apr;135(4):837-42. doi: 10.1016/j.jtcvs.2007.11.011. PMID 18374764
- [Background] Iyoda A, Baba M, Shibuya K, Moriya Y, Yasufuku K, Sekine Y, Iizasa T, Hiroshima K, Nakatani Y, Fujisawa T. Transbronchial fine needle aspiration cytological examination: a useful tool for diagnosing primary lung cancer. Thorac Cardiovasc Surg. 2006 Mar;54(2):117-9. doi: 10.1055/s-2005-865924. PMID 16541353
- [Background] Roth K, Hardie JA, Andreassen AH, Leh F, Eagan TM. Predictors of diagnostic yield in bronchoscopy: a retrospective cohort study comparing different combinations of sampling techniques. BMC Pulm Med. 2008 Jan 26;8:2. doi: 10.1186/1471-2466-8-2. PMID 18221551
- [Background] Mondoni M, Sotgiu G, Bonifazi M, Dore S, Parazzini EM, Carlucci P, Gasparini S, Centanni S. Transbronchial needle aspiration in peripheral pulmonary lesions: a systematic review and meta-analysis. Eur Respir J. 2016 Jul;48(1):196-204. doi: 10.1183/13993003.00051-2016. Epub 2016 May 12. PMID 27174878
- [Background] Oki M, Saka H, Ando M, Asano F, Kurimoto N, Morita K, Kitagawa C, Kogure Y, Miyazawa T. Ultrathin Bronchoscopy with Multimodal Devices for Peripheral Pulmonary Lesions. A Randomized Trial. Am J Respir Crit Care Med. 2015 Aug 15;192(4):468-76. doi: 10.1164/rccm.201502-0205OC. PMID 26039792
- [Background] Gasparini S. It is time for this 'ROSE' to flower. Respiration. 2005 Mar-Apr;72(2):129-31. doi: 10.1159/000084041. No abstract available. PMID 15824520
- [Background] Gasparini S, Zuccatosta L, De Nictolis M. Transbronchial needle aspiration of mediastinal lesions. Monaldi Arch Chest Dis. 2000 Feb;55(1):29-32. No abstract available. PMID 10786422
- [Background] Gasparini S. GPS may help drivers reach their destination, but the capability to drive a car is still necessary. Traditional and technology-guided transbronchial needle aspiration. Respiration. 2007;74(4):379-81. doi: 10.1159/000103206. No abstract available. PMID 17641483
- [Background] Gasparini S. Evolving role of interventional pulmonology in the interdisciplinary approach to the staging and management of lung cancer: bronchoscopic mediastinal staging of lung cancer. Clin Lung Cancer. 2006 Sep;8(2):110-5. doi: 10.3816/CLC.2006.n.038. PMID 17026811